CLINICAL TRIAL: NCT04448444
Title: Brain Activity Changes Following Neuroproprioceptive Physiotherapy in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-VP/22/0/2014/2
Record Dates: First submitted 2020-06-18; First posted 2020-06-25 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Neuronal Plasticity; Multiple Sclerosis; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study was designed as parallel group (outpatients) randomized comparison of two kinds of physiotherapeutic interventions referred to healthy controls.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Program Activating Therapy (MPAT) (Experimental): The MPAT was chosen for our clinical experience - it was developed and verified by our team. In this therapy, patients are corrected into a postural position where the joints are functionally centred. Then somatosensory (manual and verbal) stimuli are applied to activate motor programs in the brain, which then lead to the co-contraction of the patient's whole body when the patient is lying, sitting, standing up or moving forward. Activated programs are repeated under various conditions and in different situations and environments to teach the patients to use the acquired motor skills automatically in daily life.
  Interventions: Behavioral: Motor Program Activating Therapy
- Vojta Reflex Locomotion (VRL) (Experimental): VRL was developed by prof. Vojta and is standardly used in the Czech Republic. In this therapy, patients should be set up into the precisely given initial position with defined angular setting of extremities. In each position (supine, prone, lying on the side, and low kneeling position), activation points (zones) are stimulated with precise localization and pressure direction. Such stimulation activates one of the global movement patterns (reflex turning and reflex creeping) corresponding to the initial position. In addition to motor involuntarily reaction, also sensory and autonomic response is activated.
  Interventions: Behavioral: Vojta reflex locomotion
- healthy controls (No Intervention): sex and age matched healthy controls

INTERVENTIONS:
Behavioral: Motor Program Activating Therapy — Patients undergo ambulatory physiotherapy - Motor Program Activating Therapy (2 months, twice a week, 1 hour of duration). Therapy was undertaken at the ambulatory section of the Department of Neurology, Kralovske Vinohrady University Hospital in Prague.
  Arms: Motor Program Activating Therapy (MPAT)
Behavioral: Vojta reflex locomotion — Patients undergo ambulatory physiotherapy - Vojta Reflex Locomotion Therapy (2 months, twice a week, 1 hour of duration). Therapy was undertaken at the Department of Rehabilitation and Sport Medicine, Motol University Hospital.
  Arms: Vojta Reflex Locomotion (VRL)

SUMMARY:
Imaging methods bring new possibilities for describing the brain plasticity processes that underly the improvement of clinical function after physiotherapy in people with multiple sclerosis (pwMS). The study determined whether facilitation physiotherapy could enhance brain plasticity, compared two facilitation methods, and looked for any relation to clinical improvement in pwMS.

DETAILED DESCRIPTION:
The study was designed as parallel group randomized comparison of two kinds of physiotherapeutic interventions referred to healthy controls.

MS patients were examined by fMRI (primary outcomes) and clinical tests (secondary outcomes) at the beginning of study. Then, they were randomly divided into two groups (by drawing lots in a 1:1 ratio). The first group underwent Vojta reflex locomotion (VRL), and the second Motor Program Activating Physiotherapy (MPAT). The length and intensity of treatment was the same in both groups (two months, one hour twice a week). After the treatment, a clinical and fMRI examination was performed. Healthy volunteers underwent an fMRI examination that was considered to be a control.

ELIGIBILITY:
Inclusion Criteria:

* definite MS
* stable clinical status in the preceding 3 months
* imuno-modulatory treatment for at least two years (including glatiramer acetate, interferon beta-1a, 1b, mitoxantrone, fingolimod, natulizumab)
* Expanded Disability Status Scale (EDSS)≤6
* predominant motor impartment
* six months or more without any physiotherapy
* ability to undergo ambulatory physiotherapy

Exlusion criteria:

-other neurological disease or conditions disabling movement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Brain activity | 0 month
  fMRI examinations on 3T magnetic resonance scanner (Siemens Trio Tim, Erlangen, Germany) using a 12-channel head coil (different pattern of brain activity in healthy and people with MS)
Brain activity | 0 and 2 months
  fMRI examinations on 3T magnetic resonance scanner (Siemens Trio Tim, Erlangen, Germany) using a 12-channel head coil (different pattern of brain activity before and after two months of physiotherapeutic program)

SECONDARY OUTCOMES:
Nine Hole Peg Test - NHPT | 2 months
  measure finger dexterity (quicker time means better function)
Paced Auditory Serial Addition Test - PASAT | 2 months
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio record to ensure standardization in the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The score for the PASAT is the total number correct out of 60 possible answers.
Berg Balance Scale - BBS | 2 months
  14 items objective measure of static balance and risk of falls (0 the best, 56 the worse)
Timed 25 Foot Walk - T25FW | 2 months
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. The score for the T25-FW is the average of the two completed trials.
Timed Up and Go - TUG | 2 months
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, Ph.D., Principal Investigator — Charles University, Czech Republic